CLINICAL TRIAL: NCT02019030
Title: Treatment of Symptomatic BPH Patients Undergoing Anticoagulant Therapy Using the PlasmaButton Vaporization Electrode - An Observational Study
Brief Title: Treatment of Symptomatic BPH Patients Undergoing Anticoagulant Therapy Using the PlasmaButton Vaporization Electrode
Status: Terminated | Type: Observational
Why Stopped: Not meeting enrollment goals
Sponsor: Olympus Corporation of the Americas (Industry)
Collaborators: Loma Linda University (Other); VA Greater Los Angeles Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 5130322
Record Dates: First submitted 2013-12-11; First posted 2013-12-24 (Estimated); Last update posted 2018-04-04 (Actual); Status verified 2018-04

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: benign prostatic hyperplasia; Transurethral vaporization of prostate
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- BPH on anticoagulation: Patients with Benign Prostatic Hyperplasia (BPH) undergoing Transurethral Vaporization of Prostate and are on anticoagulant medication

SUMMARY:
The purpose of this observational study is to evaluate the outcomes of using the PlasmaButton electrode in the treatment on Benign Prostatic Hyperplasia (BPH) while on anticoagulation medication.

ELIGIBILITY:
Inclusion Criteria:

* Men with obstructive symptoms due to benign prostatic hyperplasia who are also on anticoagulant regimen.
* Anticoagulant regiments include: Aspirin 81mg, Aspirin 325mg, Adenosine diphosphate (ADP) receptor inhibitors, Cilostazol, Dabigatran, Dipyridamole, or Warfarin. The patient will be stable on their dosage regimen for at least 3 months.
* Maximum flow rate <15ml/s by uroflowmetry.
* International Prostate Symptom Score (IPSS)≥10.

Exclusion Criteria:

* Patients with coagulopathy, INR exceeding 3.
* Anti-coagulation dose changes within 3 months of surgery.
* Patients not medically cleared to undergo surgery for medical reasons.
* Patients with neurogenic bladder (bladder affected due to a neurologic cause).
* Urethral stricture, obstruction due to stricture.
* Suspected bladder or prostate cancer.
* Prostate size greater than 80 cc.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Symptomatic BPH patients seen at Urology clinic at Loma Linda University Medical Center and VA Greater Los Angeles Healthcare System
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2017-01-03 (Actual); Study Completion 2017-01-03 (Actual)

PRIMARY OUTCOMES:
Complication rates when the PlasmaButton Electrode is used to perform TUVP (Transurethral Vaporization of the Prostate) on patients on anticoagulants | Introperative

SECONDARY OUTCOMES:
Assessment of subjective patient improvement on the International Prostate Symptom Score questionnaire | Before surgery and 1, 3, 6 month follow up visits
Assessment of subjective patient improvement on the Sexual Health Inventory for Men (SHIM) score | Before surgery and 1, 3, 6 month follow-up
Measurement of maximum urine flow rate as measured by urine flowmetry | Before surgery and 1, 3, 6 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Edmund Ko, MD, Principal Investigator — Loma Linda University Medical Center; Carol J Bennett, MD, Principal Investigator — VA Greater Los Angeles Healthcare System
Locations (2):
- United States (2):
  - Loma Linda University Medical Center Urology Department, Loma Linda, California
  - VA Greater Los Angeles Healthcare System, Los Angeles, California